CLINICAL TRIAL: NCT00241254
Title: A Double-blind, Two-arm, Multicenter, Randomized Trial to Evaluate Efficacy of Cyclophosphamide Versus Methylprednisolone in Patients With Recent Secondary Progressive Multiple Sclerosis: P.R.OM.E.S.S Study
Brief Title: Efficacy of Cyclophosphamide Versus Methylprednisolone in Patients With Secondary Progressive Multiple Sclerosis
Acronym: PROMESS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9408-04; 2004-005
Record Dates: First submitted 2005-10-17; First posted 2005-10-18 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Multiple Sclerosis, Chronic Progressive
Keywords: Multiple Sclerosis, Chronic Progressive; Cyclophosphamide; Methylprednisolone; Randomized Controlled Trials; Double-Blind Study
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — Cyclophosphamide; Pharmaceutical Preparations; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Cyclophosphamide
  Interventions: Drug: Cyclophosphamide (drug)
- 2 (Active Comparator): Methylprednisolone
  Interventions: Drug: Methylprednisolone (drug)

INTERVENTIONS:
Drug: Cyclophosphamide (drug) — IV cyclophosphamide infusion administered every 4 weeks during 1 year and every 8 weeks during 1 year.
  Arms: 1
Drug: Methylprednisolone (drug) — Control group : IV methylprednisolone infusion administered every 4 weeks during 1 year and every 8 weeks during 1 year.
  Arms: 2

SUMMARY:
Preliminary not-controlled clinical studies of the efficacy of monthly intravenous cyclophosphamide administration in secondary progressive multiple sclerosis reported encouraging results, but no randomized controlled trial has been conducted so far. The primary objective of this trial is to evaluate the efficacy of IV cyclophosphamide as compared to IV methylprednisolone administered every 4 weeks during 1 year and every 8 weeks during 1 year, on the delay to confirmed disability deterioration as assessed by the Expanded Disability Status Scale (EDSS) in patients with secondary progressive multiple sclerosis. The secondary objectives are to evaluate safety, tolerability and efficacy at 2 years on the Multiple Sclerosis Functional Composite (MSFC), the percentage of patients with disability deterioration (EDSS) and the number of relapses. An intention-to-treat statistical analysis will be carried out.

DETAILED DESCRIPTION:
Background

Preliminary not-controlled clinical studies of the efficacy of monthly intravenous cyclophosphamide administration in secondary progressive multiple sclerosis reported encouraging results, but no randomized controlled trial has been conducted so far. A slight efficacy of Methylprednisolone has been reported in this indication.

Objectives

The primary objective is to evaluate the efficacy of IV cyclophosphamide on the prevention of disability deterioration in patients with secondary progressive multiple sclerosis.

The secondary objectives are to evaluate safety, tolerability and efficacy of IV cyclophosphamide on the Multiple Sclerosis Functional Composite (MSFC) and the number of relapses.

Study design

Randomized double-blind two-arm controlled trial.

Intervention

Experimental group : IV cyclophosphamide infusion administered every 4 weeks during 1 year and every 8 weeks during 1 year.

Control group : IV methylprednisolone infusion administered every 4 weeks during 1 year and every 8 weeks during 1 year.

Outcomes

Primary outcome : delay to disability deterioration as assessed by the Expanded Disability Status Scale (EDSS: 0.5 or 1 point increase, depending on baseline score) evaluated every 4 weeks for one year, then every 8 weeks for one year.

Secondary outcomes : proportion of patients with disability deterioration (EDSS: 0.5 or 1 point increase, depending on baseline score), Multiple Sclerosis Functional Composite (MSFC) and the Z scores of MSFC three components, number of MS relapses, proportion of patients with adverse events and delay of occurrence of adverse events, quality of life questionnaires.

* Quality of life questionnaires
* Disability self-assessment questionnaires Main time of assessment : 2 years.

Sample size

360 patients

Statistical analysis

Intention-to-treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* Multiple sclerosis (MS) subjects (Mc Donald et al criteria),
* Aged 18 to 65
* Diagnosis of secondary progressive MS ( Lublin and Reingold criteria)
* Progressive deterioration phase of at least 6 months and less than 4 years.
* Reduction of walking capacity and increase EDSS not ascribed to consequence of relapses (at least 0.5 point) in the last 12 months
* EDSS between 4.0 and 6.5 included
* Female participating must use contraceptives while on study drug
* Written informed consent
* Patient protected by French social security system

Exclusion Criteria:

* Others diseases interfering with MS or treatment
* Recent history (within the previous 2 years) of drug or alcohol abuse.
* Patients with psychiatric illnesses who are unable to provide written, informed consent prior to any testing under this protocol
* Hemorrhagic cystitis
* Pregnant or lactating women
* Known allergy at cyclophosphamide, corticoids and in particular methylprednisolone
* Persistent infectious diseases
* Patients with bladder permanent catheterization
* Known history of cardiac arrhythmia after methylprednisolone intravenous treatment
* Abnormal screening/baseline blood tests exceeding any of the limits defined below : Hb < 9g/dl or Total white blood cell count less than 3 000/mm3 or lymphocytes count less than 900/ mm3 or Platelet count less than 125 000/mm3
* Gastric or duodenal ulcer in evolution
* Gut diverticulosis
* Diabetes mellitus
* Known history of active hepatitis (ASAT >3 X ULN)
* Known history of renal failure (creatinine level > 180 µmol/L)
* Psychosis
* Current or past (< 3 months) participation in another drug trial
* Prior use of cyclophosphamide, lymphoid irradiation, monoclonal antibodies anti CD4 or anti CD52 or anti-VLA-4 therapies, cladribine ou cyclosporine A
* Other clinical types of MS : Secondary progressive phase evolving for more than 4 years ; Remittent type of MS without progression between relapses ; Primary progressive type of MS
* Use of interferon beta, methotrexate or imurel in the month prior to study.
* Treatment with intravenous monthly corticoids in the year prior to study.
* Treatment with corticoids (3 to 5 days) in the 2 month prior to study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2005-12; Primary Completion 2010-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Delay to disability deterioration as assessed by the Expanded Disability Status Scale (EDSS: 0.5 or 1 point increase, depending on baseline score) | every 4 weeks for one year, then every 8 weeks for one year

SECONDARY OUTCOMES:
Proportion of patients with disability deterioration (EDSS: 0.5 or 1 point increase, depending on baseline score) | every month during one year then every two months during the 2nd year
Multiple Sclerosis Functional Composite (MSFC) and the Z scores of MSFC three components | Visit number 1, 2, 13(at one year),19 (at two years) and 20 (last visit)
Number of MS relapses | all along the follow up period
Proportion of patients with adverse events and delay of occurrence of adverse events | all along the follow up period
Quality of life questionnaires | visit 2, 13(at one year) and 19 (at two years)
Disability self-assessment questionnaires | visite 2, 13 et 19

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Brochet, Professor, Principal Investigator — University Hospital, Bordeaux, France; Paul Perez, Dr, Study Chair — University Hospital, Bordeaux, France
Locations (26):
- France (26):
  - CH de la Cote Basque, Bayonne
  - CHU Besançon, Besançon
  - Hôpital Pellegrin, Département de neurologie, Bordeaux
  - CHU Caen, Caen
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - AP HP Henri Mondor, Créteil
  - CHU Dijon, Dijon
  - CHU Lille Hôpital Salengro, Lille
  - CHU Limoges, Limoges
  - GHICL Hôpital St. Philibert, Lomme
  - (CHU Lyon) Hôpital neurologique, Lyon
  - Hôpital La Timone, Marseille
  - (CHR Metz-Thionville) Hôpital Notre Dame de Bon Secours, Metz
  - (CHU Montpellier), Hôpital de Gui de Chauliac, Montpellier
  - CHU Nancy Hôpital central, Nancy
  - Hôpital Guillaume et René Laënnec, Nantes
  - CHU Nice Hôpital Pasteur, Nice
  - (CHU Nîmes) Hôpital Caremeau, Nîmes
  - Fondation Rothschild, Paris
  - (AP HP) Hôpital Tenon, Paris
  - Centre Hospitalier de Pau, Pau
  - CHU de POISSY, Poissy
  - (CHU Reims) Hôpital Robert Debré, Reims
  - CHU Ponchaillou, Rennes
  - CH d'Angoulême Girac, Saint-Michel
  - (CHRU Starsbourg) Hôpital civil, Strasbourg

REFERENCES:
- [Derived] Brochet B, Deloire MS, Perez P, Loock T, Baschet L, Debouverie M, Pittion S, Ouallet JC, Clavelou P, de Seze J, Collongues N, Vermersch P, Zephir H, Castelnovo G, Labauge P, Lebrun C, Cohen M, Ruet A; PROMESS study investigators. Double-Blind Controlled Randomized Trial of Cyclophosphamide versus Methylprednisolone in Secondary Progressive Multiple Sclerosis. PLoS One. 2017 Jan 3;12(1):e0168834. doi: 10.1371/journal.pone.0168834. eCollection 2017. PMID 28045953